CLINICAL TRIAL: NCT01181076
Title: Individualized Nutrition for Adult Recipients of Allogeneic Stem Cell Transplants - Effect on Quality of Life
Acronym: NASQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, Kristin Joan Skaarud, Per Ole Iversen, MD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: S-09136c
Record Dates: First submitted 2010-08-04; First posted 2010-08-13 (Estimated); Results first posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Effect of Individualized Nutrition on Quality of Life
Keywords: Stem cell transplantation; Individualized Nutrition; Quality of life; Oral Mucositis; Adult
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Individualized Nutrition (Experimental)
  Interventions: Dietary Supplement: Individualized Nutrition
- Control group (No Intervention): The patients in the control group will be nourished after established routine, first by the oral route, later by the PN route. Naso-jejunal tube will not be inserted and enteral nutrition will not be given.

INTERVENTIONS:
Dietary Supplement: Individualized Nutrition — The patients who are able to achieve oral nutrition requirement will receive a therapeutic diet using regular foods, which is lactose-reduced and energy-enriched. The naso-jejunal tube will be inserted during the first five days after transplantation. EN will be given when oral intake discontinue. EN with an additional PN will be given if the estimated requirements by the enteral route is lower than reference values.
  Arms: Individualized Nutrition

SUMMARY:
Aim

Allogeneic stem cell transplantation (allo-SCT) combined with several cycles of intensive chemotherapy is the only curative treatment for several malignant blood diseases. Most allo-SCT patients who are treated with intensive chemotherapy often have reduced nutritional status. Several studies have evaluated the effect of different nutrition intervention for allo-SCT patients, but there have not been found evidence-based recommendations for energy requirements, use of enteral nutrition (EN) and/or parenteral nutrition (PN). We are not aware of studies using QoL as end-point among allo-SCT patients allocated to specific nutrition intervention.

Main hypothesis:

Patients who receive individualized nutrition have better "global" QoL assessed with the European Organisation for Research and Treatment in Cancer (EORTC) QLQ-HDC29 tool three months after SCT

Sub-hypotheses:

Patients who receive individualized nutrition have:

i) less often oral mucositis grade 3-4. ii) better nutrition status iii) decreased length of hospital stay, less episodes with fever, earlier engraftment and less often acute graft versus host disease (GVHD) grade 3-4, and iv) better main QoL scores on the scale for physical and social functions, fatigue, loss of appetite, nausea/vomiting and diarrhoea three months after allogeneic SCT, compared to the control group.

Patients and methods A minimum sample of 100 patients will be included in the study. The patients enrolled in the study will be randomly assigned to the intervention- or control group. The patients in the intervention group will receive a therapeutic diet in combination with tube feeding with an additional PN if the estimated requirements by the enteral route is lower than reference values. The patients in the control group will receive nutrition support after established routine, first by the oral route, later by the PN route.

DETAILED DESCRIPTION:
Patients and methods

A minimum sample of 100 patients will be included in the study. This is the result of a power calculation where a difference of 15 of global QoL is the primary end-point. All patients who fulfil the inclusion criteria and are offered allo-SCT with myeloablative condition are invited to participate in the study about 1-3 months before commencing the treatment. The patients have to give their written informed consent to participate in the study. The patients enrolled in the study will be randomly assigned in blocks to the intervention- or control group. The main end-point is three months after SCT. We will follow the patients throughout the first year after SCT.

Nutrition intervention

The interventions start when the patients are arriving at the hospital for SCT and consist of individualized nutrition supplement for each patient until discharge. The severity of nausea, vomiting, diarrhea and mouth soreness will be a measure of the administration route of nutrition (oral, PN and/or EN). The energy requirements will be calculated and the intake monitored. The energy intake will continuously be adjusted to the energy requirements. The patients who are able to achieve oral nutrition requirement will receive a therapeutic diet using regular foods, which is lactose-reduced and energy-enriched. The naso-jejunal tube will be inserted during the first five days after transplantation. EN will be given when oral intake discontinue, and an additional PN will be given if the estimated requirements by the enteral route is lower than reference values. Dislodged tubes will promptly be replaced until two times in the stomach. If the tube dislodge for more than two times, or voluminous diarrhea appears, or the patients refuse the tube, the patients will be nourished by the PN route only. The patients in the intervention group will receive dietary recommendation before leaving the hospital. The patients in the control group will be nourished after established routine, first by the oral route, later by the PN route. Naso-jejunal tube will not be inserted and enteral nutrition will not be given.

Measurement of quality of life, mucositis and nutrition status

The patients score on the EORTC QLQ-C30 form at admission, i.e. 8 days prior to SCT, then after 3 and 6 weeks and after 3, 6, 9 and 12 months. At the same time we will measure the following several markers of nutritional status and parameters of hemostasis. We will also record routine clinical parameters as well as anthropometry and body composition using electrical bioimpedance. WHO Oral Toxicity Grading Scale will be used to measure oral mucositis. In addition we will use the Patient-Generated Subjective Global Assessment (PG-SGA).

ELIGIBILITY:
Inclusion Criteria:

* acute lymphatic leukaemia, acute myeloid leukaemia, chronic myeloproliferative disease and chronic myelogenous leukaemia and other disorders accepted for allogeneic stem cell transplantation, following myeloablative conditioning

Exclusion Criteria:

* unable to give informed consent
* unable to adhere to protocol due to reasons unrelated to the hematological condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2010-08-10 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Per O Iversen, MD, Principal Investigator — Oslo University Hospital
Locations (2):
- Oslo University Hospital, Oslo, Norway
- Pavlov State Medical University of St. Petersburg, Saint Petersburg, Russia

REFERENCES:
- [Derived] Gudmundstuen AM, Iversen PO, Pesonen M, Hjermstad MJ, Bye A, Tjonnfjord GE, Skaarud KJ. Comparing indirect calorimetry and predictive equations for energy expenditure - 1 year follow-up of adult hematopoietic stem cell transplanted recipients. Clin Nutr ESPEN. 2025 Dec;70:218-226. doi: 10.1016/j.clnesp.2025.09.027. Epub 2025 Sep 30. PMID 41038512
- [Derived] Skaarud KJ, Gudmundstuen AM, Pesonen M, Hjermstad MJ, Iversen PO, Tjonnfjord GE. The role of fat-soluble vitamins for graft-versus host disease after myeloablative conditioning in allogeneic stem cell transplanted patients. Sci Rep. 2025 Jan 11;15(1):1675. doi: 10.1038/s41598-024-84805-2. PMID 39799129
- [Derived] Skaarud KJ, Hov JR, Hansen SH, Kummen M, Valeur J, Seljeflot I, Bye A, Paulsen V, Lundin KEA, Troseid M, Tjonnfjord GE, Iversen PO. Mortality and microbial diversity after allogeneic hematopoietic stem cell transplantation: secondary analysis of a randomized nutritional intervention trial. Sci Rep. 2021 Jun 2;11(1):11593. doi: 10.1038/s41598-021-90976-z. PMID 34078971

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As determined
Period: Overall Study
Arm/Group | Individualized Nutrition | Control Group
Started | 59 | 60
Completed | 40 | 48 (As determined)
Not Completed | 19 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Individualized Nutrition | Control Group | Total
Number analyzed (Participants) | 59 | 60 | 119
Age, Continuous [Median (Full Range); unit: years] | 45 [19 to 65] | 41 [18 to 62] | 42 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 25 | 45
  Male | 39 | 35 | 74
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Norway | 59 | 60 | 119

OUTCOME MEASURES:

1. Primary Outcome: Global Quality of Life Score
Description: A score for measurement of global quality of life will be obtained from the European Organisation for Research and Treatment of Cancer, form EORTC QLQ-C30. The scores range from 0 to 100, higher scores mean better outcome.
Time Frame: 3 month after transplantation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Individualized Nutrition | Control Group
Number analyzed (Participants) | 40 | 48
units on a scale | 58.8 (19.2) | 55.4 (23.3)

2. Secondary Outcome: Number of Underweight Participants
Description: Nutritional status will be assessed with anthropometry, biomarkers and bioimpedance. Here the number of underweight participants is reported.
Time Frame: 3 month after transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized Nutrition | Control Group
Number analyzed (Participants) | 59 | 60
Participants | 2 | 4

3. Secondary Outcome: Number of Episodes With Fever
Description: Fever episodes
Time Frame: Up to 8 months
Measure: Number; unit: Fever episodes
Arm/Group | Individualized Nutrition | Control Group
Number analyzed (Participants) | 59 | 60
Fever episodes | 55 | 59

4. Secondary Outcome: Duration Between Stem Cell Transplantation and Day of Engraftment.
Description: Engraftment was judged by the number of days to neutrophils ≥0.2 × 109/l.
Time Frame: Up to 1 months
Measure: Median (Full Range); unit: days
Arm/Group | Individualized Nutrition | Control Group
Number analyzed (Participants) | 59 | 60
days | 15 [11 to 31] | 16 [10 to 30]

5. Secondary Outcome: Frequency of Acute Graft Versus Host Disease Grade 3-4
Time Frame: Up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized Nutrition | Control Group
Number analyzed (Participants) | 59 | 60
Participants | 7 | 13

6. Secondary Outcome: Number of Participants With Hospital Stay
Time Frame: Up to 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized Nutrition | Control Group
Number analyzed (Participants) | 59 | 60
Participants | 37 | 39

7. Secondary Outcome: Number of Participants With Pain, as Determined by EORTC QLQ C30
Description: These scores (range 0-100) will be assessed with the EORTC QLQ C30 form. Higher scores means more pain.
Time Frame: 3 months after transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized Nutrition | Control Group
Number analyzed (Participants) | 59 | 60
Participants | 40 | 48

8. Secondary Outcome: Number of Participants With Oral Mucositis Grade 3-4
Description: Oral mucositis will be graded according to the World Health Organization Oral Toxicity Grading Scale, range 0-4 in scores, higher scores mean worse outcome.
Time Frame: Up to 3 months
Measure: Number; unit: participants
Arm/Group | Individualized Nutrition | Control Group
Number analyzed (Participants) | 59 | 60
participants | 42 | 45

ADVERSE EVENTS:
Time Frame: 6 years
Arm/Group | Individualized Nutrition | Control Group
All-Cause Mortality (participants affected / at risk) | 9/59 | 5/60
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/60
Other Adverse Events (participants affected / at risk) | 0/59 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2009-10-23): https://cdn.clinicaltrials.gov/large-docs/76/NCT01181076/Prot_000.pdf